CLINICAL TRIAL: NCT00311792
Title: Transfer of Skills From LapSimGyn VR-Simulator to a Laparoscopic Salpingectomy
Brief Title: Transfer of Skills From VR-Trainer to Operation Room
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KF 01283756; 959587647
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: Clinical Competence
Keywords: training; teaching; curriculum

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Simulator training
  Interventions: Behavioral: LapSimGyn training until expert proficiency level is reached
- 2 (Active Comparator): Traditional Clinical education at operating room
  Interventions: Behavioral: Traditional clinical education

INTERVENTIONS:
Behavioral: LapSimGyn training until expert proficiency level is reached — Two consecutive simulations reaching predefined expert level
  Arms: 1
Behavioral: Traditional clinical education
  Arms: 2

SUMMARY:
The purpose is to determine if skills obtained by training in the laparoscopic virtual reality simulator LapSimGyn can be transferred to a real laparoscopic operation measured as improved score in a technical skills assessment.

DETAILED DESCRIPTION:
The purpose is to determine if skills obtained by training in the laparoscopic virtual reality simulator LapSimGyn can be transferred to a real laparoscopic operation measured as improved score in a technical skills assessment. Design: prospective randomized double blinded intervention study.

Subjects:Younger gynaecologists (Postgraduate year 2-8) Half are having conventional training the other half is undergoing virtual reality simulator training before performing their first laparoscopic salpingectomy.

Outcome is measured by blinded video evaluation with criteria. The criteria is defined in the previous validated scoring system Objective Structured Assessment of Technical Skills (OSATS)

ELIGIBILITY:
Inclusion Criteria:

* Gyn/obs trainee 1.-2. year, with no experience from advanced laparoscopy

Exclusion Criteria:

* Advanced laparoscopic experience
* Previous training in simulator

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Rating Scale Score | 1 day

SECONDARY OUTCOMES:
Time used to perform operation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bent Ottesen, MD Dr.Sci, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Issenberg SB, McGaghie WC, Petrusa ER, Lee Gordon D, Scalese RJ. Features and uses of high-fidelity medical simulations that lead to effective learning: a BEME systematic review. Med Teach. 2005 Jan;27(1):10-28. doi: 10.1080/01421590500046924. PMID 16147767
- [Derived] Larsen CR, Soerensen JL, Grantcharov TP, Dalsgaard T, Schouenborg L, Ottosen C, Schroeder TV, Ottesen BS. Effect of virtual reality training on laparoscopic surgery: randomised controlled trial. BMJ. 2009 May 14;338:b1802. doi: 10.1136/bmj.b1802. PMID 19443914